CLINICAL TRIAL: NCT02030704
Title: Comprehensive 'Bio-Imaging' Using Quantitative Coronary Plaque Composition Assessment and the High-sensitive Troponin T for the Prediction of Cardiac Outcomes.
Brief Title: CCTA-based Coronary Plaque Characterization and High-sensitive Troponin T for the Prediction of Cardiovascular Outcomes
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Semmelweis University Heart and Vascular Center (Other); Heidelberg University (Other)
Responsible Party: Principal Investigator, GKorosoglou, Prof. Dr. med., University Hospital Heidelberg
Other Study IDs: HDCCTA01
Record Dates: First submitted 2014-01-07; First posted 2014-01-08 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Coronary Artery Disease; Noninvasive Plaque Characterization
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Atherosclerotic Plaque

SUMMARY:
To determine the ability of semi-automated plaque assessment in cardiac computed tomography angiography (CCTA) and high sensitive troponin T (hsTnT) for the risk stratification of patients at intermediate risk for coronary artery disease (CAD).

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for CCTA according to the current appropriate use criteria

Exclusion Criteria:

* non-sinus rhythm
* acute coronary syndromes
* cardiomyopathies
* moderate or severe valvular disease
* elevated serum creatinine (>1.5 mg/dl)
* history or ECG signs of previous myocardial infarction
* severe iodine allergy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients scheduled to undergo CCTA
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2008-02; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Cardiac death | two years
Nonfatal myocardial infarction | two years

SECONDARY OUTCOMES:
Myocardial revascularization including PCI and CABG | two years
  PCI - Percutaneous Coronary Intervention CABG - Coronary Artery Bypass Grafting

CONTACTS AND LOCATIONS:
Overall Officials: Grigorios Korosoglou, Prof. Dr. med., Principal Investigator — University of Heidelberg, Department of Cardiology, Heidelberg, Germany.
Locations (2):
- University of Heidelberg, Department of Cardiology, Heidelberg, Baden-Wurttemberg, Germany
- MTA-SE Lendület Cardiovascular Imaging Research Group, Heart and Vascular Center, Semmelweis University, Budapest, Hungary

REFERENCES:
- [Background] Korosoglou G, Mueller D, Lehrke S, Steen H, Hosch W, Heye T, Kauczor HU, Giannitsis E, Katus HA. Quantitative assessment of stenosis severity and atherosclerotic plaque composition using 256-slice computed tomography. Eur Radiol. 2010 Aug;20(8):1841-50. doi: 10.1007/s00330-010-1753-3. Epub 2010 Mar 20. PMID 20306078